CLINICAL TRIAL: NCT00854607
Title: A Prospective, Non-Intervention, Observational Assessment of the Correlation Between Circulating Biomarkers of Fungal Bioburden and Clinical Outcome in the Setting of Invasive Aspergillosis
Brief Title: An Observational Study of Fungal Biomarkers (MK-0000-089)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-089; 2009_553 (Other: Merck)
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Aspergillosis
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected for 12 weeks to evaluate levels of fungal biomarkers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Invasive Aspergillosis: Observational
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Blood samples will be collected for 12 weeks to evaluate levels of fungal biomarkers.

SUMMARY:
The purpose of this study is to evaluate the relationship between fungal biomarker levels during anti-fungal therapy and the success of treatment for fungal infection. The primary hypothesis is that over the initial two weeks of anti-fungal therapy, fungal biomarkers from participants with invasive aspergillosis (IA) will be lower for those with a successful clinical outcome compared to those with a failed clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Is 16 years of age or older
* Female is either post-menopausal, surgically sterilized, willing to use 2 adequate methods of birth control, or agrees to abstain from heterosexual activity throughout the study
* Female of child bearing potential must have a negative pregnancy test
* Male is surgically sterilized, agrees to use an adequate method of contraception, or agrees to abstain from heterosexual activity for the duration of the study
* Has possible, probable, or confirmed invasive aspergillosis (IA)
* Has had a computed tomography (CT) or magnetic resonance imaging (MRI) scan 72 hours prior to initiation of anti-fungal therapy

Exclusion Criteria:

* Has had hemodialysis using cellulose membrane within 2 weeks of study start

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected through collaborations with clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Neofytos D, Railkar R, Mullane KM, Fredricks DN, Granwehr B, Marr KA, Almyroudis NG, Kontoyiannis DP, Maertens J, Fox R, Douglas C, Iannone R, Kauh E, Shire N. Correlation between Circulating Fungal Biomarkers and Clinical Outcome in Invasive Aspergillosis. PLoS One. 2015 Jun 24;10(6):e0129022. doi: 10.1371/journal.pone.0129022. eCollection 2015. PMID 26107507

RESULTS

PARTICIPANT FLOW:
Groups:
- Invasive Aspergillosis: Participants who enrolled with a presumptive diagnosis of possible, probable or proven Invasive Aspergillosis (IA) infection, were started on standard of care antifungal therapy. Within 14 days of the start of therapy participants were re-evaluated, and those diagnosed with possible IA were discontinued from the study, while those with probable and proven IA were defined as the baseline population
Period: Enrollment
Arm/Group | Invasive Aspergillosis
Started | 116
Completed | 116
Not Completed | 0
Period: 2 Weeks After Start Anti-fungal Therapy
Arm/Group | Invasive Aspergillosis
Started | 116
Completed | 51
Not Completed | 65
Not completed — Diagnosed with Possible IA | 65

BASELINE CHARACTERISTICS:
Groups:
- Invasive Aspergillosis: Participants who enrolled with a presumptive diagnosis of possible, probable or proven IA infection, were started on standard of care antifungal therapy. Within 14 days of the start of therapy participants were re-evaluated, and those diagnosed with possible IA were discontinued from the study, while those with probable and proven IA were defined as the baseline population
Arm/Group | Invasive Aspergillosis
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Average of the Z-scores of the Time-Weighted Averages (TWA) of Fungal Biomarkers Galactomannan (GM) and (1,3)-β-D-glucan (βDG) Over the First Two Weeks of Treatment for Responders (R) and Non-Responders (NonR) to Anti-fungal Treatment at Week 6.
Description: After enrollment blood was collected at baseline, twice per week for the first six weeks, then weekly through twelve weeks for biomarker analysis of GM and βDG. Clinical outcome was assessed for qualified participants at 6 and 12 weeks after initiation of antifungal treatment. For a given biomarker the Z-score is the difference from the mean of each individual TWA divided by the overall standard deviation (SD). The average of the Z-scores of the TWA for qualified participants is then calculated across all biomarkers, and used to derive the mean for R and NonR to antifungal therapy.
Time Frame: Weeks 1 and 2
Population: Surviving participants with proven or probable IA at Day 14 post antifungal therapy, who had at least two valid results for each biomarker, and whose clinical outcome was determined at Week 6.
Measure: Mean (Standard Deviation); unit: Average Z-Score
Groups:
- Non-Responders: Participants started on standard of care anti-fungal therapy on Day 0 who were diagnosed as Non-Responders at Week 6.
- Responders: Participants started on standard of care anti-fungal therapy on Day 0 who were diagnosed as Responders at Week 6.
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | 0.20 (1.32) | -0.09 (0.61)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.166, t-test, 1 sided — One-Sided P-value; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [-0.20 to 0.77]

2. Secondary Outcome: Average of the Z-scores of the Slopes of Least-Squares Straight Lines (SLSSL) Fitted to the Fungal Biomarkers GM and βDG Over the First Two Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 6.
Description: After enrollment blood was collected at baseline, twice per week for the first six weeks, then weekly through twelve weeks for analysis of biomarkers GM and βDG. Clinical outcome was assessed for qualified participants at 6 and 12 weeks after initiation of antifungal treatment. For a given biomarker the Z-score is the difference from the mean of each individual SLSSL divided by the overall SD. The average Z-scores of the SLSSL for qualified participants is then calculated across all biomarkers, and used to derive the mean for R and NonR to antifungal therapy.
Time Frame: Weeks 1 and 2
Population: Surviving participants with proven or probable IA at Day 14 post antifungal therapy, who had at least two valid results for each biomarker, and had a clinical outcome determined at Week 6.
Measure: Mean (Standard Deviation); unit: Average Z-Score
Groups:
- Non-Responders: Participants started on standard of care antifungal therapy on Day 0 who were diagnosed as Non-Responders at Week 6.
- Responders: Participants started on standard of care antifungal therapy on Day 0 who were diagnosed as Responders at Week 6.
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | -0.09 (1.37) | 0.08 (0.32)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.269, t-test, 1 sided — One-Sided P-value; Mean Difference (Final Values) = -0.17, 90% CI 2-sided [-0.65 to 0.30]

3. Secondary Outcome: Average of the Z-scores of the TWA of the Changes From Baseline (CFB) of Fungal Biomarkers GM and βDG Over the First Two Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 6.
Description: After enrollment blood was collected at baseline, twice per week for the first six weeks, then weekly through twelve weeks for analysis of GM and βDG. Clinical outcome was assessed for qualified participants at 6 and 12 weeks after initiation of antifungal treatment. For a given biomarker the Z-score is the difference from the mean of each individual TWA CFB divided by the overall SD. The average of the Z-scores of the TWA CFB for qualified participants is then calculated across all biomarkers, and used to derive the mean for R and NonR to antifungal therapy.
Time Frame: Weeks 1 and 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | 0.07 (0.26) | -0.12 (0.69)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.101, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.19, 90% CI 2-sided [-0.06 to 0.44]

4. Secondary Outcome: Average of the Z-scores of the Percent Changes From Baseline (%CFB) of Fungal Biomarkers GM and βDG Over the First Two Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 6.
Description: After enrollment blood was collected at baseline, twice per week for the first six weeks, then weekly through twelve weeks for biomarker analysis of GM and βDG. Clinical outcome was assessed for qualified participants at 6 and 12 weeks after initiation of antifungal treatment. For a given biomarker the Z-score is the difference from the mean of each individual %CFB divided by the overall SD. The average of the Z-scores of the %CFB for qualified participants is then calculated across all biomarkers, and used to derive the mean for R and NonR to antifungal therapy.
Time Frame: Weeks 1 and 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | 0.02 (1.06) | -0.00 (0.79)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference Between Non-Responders and Responders; Test type: Superiority or Other; p = 0.457, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.42 to 0.47]

5. Secondary Outcome: Average of the Z-scores of the SLSSL Fitted to the Fungal Biomarkers GM and βDG Over the First Two Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 12.
Description: After enrollment blood was collected at baseline, twice per week for the first six weeks, then weekly through twelve weeks for biomarker analysis of GM and βDG. Clinical outcome was assessed for qualified participants at 6 and 12 weeks after initiation of antifungal treatment. For a given biomarker the Z-score is the difference from the mean of each individual SLSSL divided by the overall SD. The average Z-scores of the SLSSL for qualified participants is then calculated across all biomarkers, and used to derive the mean for R and NonR to antifungal therapy.
Time Frame: Weeks 1 and 2
Population: Surviving participants with proven or probable IA at Day 14 post antifungal therapy, who had at least two valid results for each biomarker, and had a clinical outcome determined at Week 12.
Measure: Mean (Standard Deviation); unit: Average Z-Score
Groups:
- Non-Responders: Participants started on standard of care anti-fungal therapy on Day 0 who were diagnosed as Non-Responders at Week 12.
- Responders: Participants started on standard of care anti-fungal therapy on Day 0 who were diagnosed as Responders at Week 12.
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 16 | 28
Average Z-Score | -0.24 (1.71) | 0.08 (0.30)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.168, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = -0.32, 90% CI 2-sided [-0.87 to 0.23]

6. Secondary Outcome: Average of the Z-scores of the TWA of the CFB of Fungal Biomarkers GM and βDG Over the First Two Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 12.
Description: as for outcome 3
Time Frame: Weeks 1 and 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 16 | 28
Average Z-Score | 0.10 (0.30) | -0.09 (0.61)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.127, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.19, 90% CI 2-sided [-0.09 to 0.46]

7. Secondary Outcome: Average of the Z-scores of %CFB of Fungal Biomarkers GM and βDG Over the First Two Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 12.
Description: as for outcome 4
Time Frame: Weeks 1 and 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 16 | 28
Average Z-Score | 0.31 (1.40) | -0.16 (0.46)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.054, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.47, 90% CI 2-sided [-0.01 to 0.96]

8. Secondary Outcome: Average of the Z-scores of the TWA of Fungal Biomarkers GM and βDG Over the First Week of Treatment for R and NonR to Anti-fungal Treatment at Week 6.
Description: After enrollment blood was collected at baseline, twice per week for the first six weeks, then weekly through twelve weeks for analysis of GM and βDG. Clinical outcome was assessed for qualified participants at 6 and 12 weeks after initiation of antifungal treatment. For a given biomarker the Z-score is the difference from the mean of each individual TWA divided by the overall SD. The average of the Z-scores of the TWA for qualified participants is then calculated across all biomarkers, and used to derive the mean for R and NonR to antifungal therapy.
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | 0.25 (1.40) | 0.04 (1.20)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.285, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.21, 90% CI 2-sided [-0.41 to 0.83]

9. Secondary Outcome: Average of the Z-scores of the TWA of Fungal Biomarkers GM and βDG Over the First Week of Treatment for R and NonR to Anti-fungal Treatment at Week 12.
Description: as for outcome 8
Time Frame: Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Average Z-Score
Groups:
- Non-Responders: Participants started on standard of care antifungal therapy on Day 0 who were diagnosed as Non-Responders at Week 12.
- Responders: Participants started on standard of care antifungal therapy on Day 0 who were diagnosed as Responders at Week 12.
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 16 | 28
Average Z-Score | 0.41 (1.61) | 0.01 (1.06)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.159, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.41, 90% CI 2-sided [-0.27 to 1.08]

10. Secondary Outcome: Average of the Z-scores of the SLSSL Fitted to the Fungal Biomarkers GM and βDG Over the First Week of Treatment for R and NonR to Anti-fungal Treatment at Week 6.
Description: as for outcome 2
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | 0.05 (0.14) | -0.10 (0.49)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.071, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.15, 90% CI 2-sided [-0.02 to 0.32]

11. Secondary Outcome: Average of the Z-scores of the SLSSL Fitted to the Fungal Biomarkers GM and βDG Over the First Week of Treatment for R and NonR to Anti-fungal Treatment at Week 12.
Description: as for outcome 2
Time Frame: Week 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 16 | 28
Average Z-Score | 0.08 (0.17) | -0.10 (0.47)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.078, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.17, 90% CI 2-sided [-0.03 to 0.38]

12. Secondary Outcome: Average of the Z-scores of the TWA of Fungal Biomarkers GM and βDG Over the First 6 Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 6.
Description: as for outcome 8
Time Frame: Weeks 1 through 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | 0.27 (1.53) | -0.12 (0.33)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.109, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.39, 90% CI 2-sided [-0.13 to 0.91]

13. Secondary Outcome: Average of the Z-scores of the TWA of Fungal Biomarkers GM and βDG Over the First 6 Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 12.
Description: as for outcome 8
Time Frame: Weeks 1 through 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 16 | 28
Average Z-Score | 0.49 (1.75) | -0.16 (0.30)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.030, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = 0.65, 90% CI 2-sided [0.09 to 1.22]

14. Secondary Outcome: Average of the Z-scores of the SLSSL Fitted to the Fungal Biomarkers GM and βDG Over the First 6 Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 6.
Description: as for outcome 2
Time Frame: Weeks 1 through 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 25 | 25
Average Z-Score | -0.08 (1.40) | 0.08 (0.21)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.293, t-test, 1 sided — One-Sided P-value; Mean Difference (Final Values) = -0.16, 90% CI 2-sided [-0.63 to 0.32]

15. Secondary Outcome: Average of the Z-scores of the SLSSL Fitted to the Fungal Biomarkers GM and βDG Over the First 6 Weeks of Treatment for R and NonR to Anti-fungal Treatment at Week 12.
Description: as for outcome 2
Time Frame: Weeks 1 through 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Average Z-Score
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 16 | 28
Average Z-Score | -0.19 (1.76) | 0.08 (0.20)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Mean Difference between Non-Responders and Responders; Test type: Superiority or Other; p = 0.213, t-test, 1 sided — One-Sided P-Value; Mean Difference (Final Values) = -0.27, 90% CI 2-sided [-0.83 to 0.29]

ADVERSE EVENTS:
Description: All enrolled participants
Groups:
- Invasive Aspergillosis: Participants who enrolled with a presumptive diagnosis of possible, probable or proven IA infection, and were started on standard of care antifungal therapy.
Arm/Group | Invasive Aspergillosis
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.